CLINICAL TRIAL: NCT05153473
Title: Retro-prospective and Observational Study of 120 Patients for the Assessment of the Safety and the Performance of the SAGITTA EVL R Stems in Hip Arthroplasties
Brief Title: Assessment of the Safety and the Performance of the SAGITTA EVL R Stems in Hip Arthroplasties
Status: Completed | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-06-EVLR-N
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2022-09

CONDITIONS: Hip Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

INTERVENTIONS:
Device: Total Hip Arthroplasty Revision — Hip revision surgery is performed to repair an artificial hip joint (prosthesis) that has been damaged over time due to an infection, or due to normal wear and tear of the prosthetic hip. Revision surgery helps to correct the problem so the hip can function normally again.

SUMMARY:
Total hip arthroplasty is the preferred treatment for hip disease (primary or secondary osteoarthritis, osteonecrosis, for example) and femoral neck fractures. Revision risk factors reported when considering the main surgical approaches. Studied from the Dutch arthroplasty registry found a revision rate in hemiarthroplasty (HA) of 1.6% at 1 year and 2.5% at 5 years postoperatively. For total hip replacement (THA), the rate was 2.4% at 1 and 4.3% at 5 years postoperatively. Analyze shows that the risk factors for hemiarthroplasty were male sex, age under 80 (regardless of gender), posterolateral approach and uncemented fixation. The risk factors for HAT were exactly the same, but they found that smoking also played a role. It should be noted that age as a risk factor for revision is not a risk during the first year after the fracture, but becomes one in the years that follow.

In order to maintain compliance with the directive on medical devices (93/42 / EEC [M5]) and the future regulation (EU) (2017/745) relating to medical devices, SERF has set up post-market clinical follow-ups ( PMCF). This PMCF study aims to improve knowledge related to the performance, safety and benefit / risk ratio of the Sagitta EVL-R stem and to monitor patient care strategy through this clinical evaluation. Significant clinical results as well as safety must be confirmed with this patient cohort. It is important to note that this cohort reflects the specific care strategy of the University Hospital of Poitiers. Therefore, the strategy could be different between hospitals and countries.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old.
* Patients that were treated with the sagitta EVL-R stem for an indication of arthroplasty and according to the Instruction For Use (IFU).
* Primary or secondary arthrosis,
* Advanced joint destruction resulting from rheumatoid arthritis or traumatic arthritis,
* A fracture or an avascular necrosis,
* Following a previous surgical operation, on condition that the new device does not interfere with the material in place.
* indicated in the case of primary or secondary arthrosis, displaced sub-capital or transcervical fracture as well as stages I and IIB bone loss according to the PAPROWSKI classification.
* The SAGITTA EVOLUTION for REVISION implant is recommended for indications according to the bone loss classifications of SOFCOT stages I to VI, PAPROSKY types I to VI and the AAOS types Ia to Ic.
* Dysplasia

Exclusion Criteria:

* Patient presenting a contraindication indicated in the IFU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment 120 adults patients representing 124 hips operated between 2011 and 2014.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Etienne GAYET, MD, Principal Investigator — Poitiers University Hospital
Locations (1):
- CHU de Poitiers, Poitiers, France

REFERENCES:
- [Background] Delaunay C, Epinette JA, Dawson J, Murray D, Jolles BM. Cross-cultural adaptations of the Oxford-12 HIP score to the French speaking population. Orthop Traumatol Surg Res. 2009 Apr;95(2):89-99. doi: 10.1016/j.otsr.2009.01.003. Epub 2009 Apr 3. PMID 19345630
- [Background] Girard J, Roche O, Wavreille G, Canovas F, Le Beguec P. Stem subsidence after total hip revision: 183 cases at 5.9 years follow-up. Orthop Traumatol Surg Res. 2011 Apr;97(2):121-6. doi: 10.1016/j.otsr.2010.10.006. Epub 2011 Mar 23. PMID 21435964
- [Background] Maradit Kremers H, Larson DR, Crowson CS, Kremers WK, Washington RE, Steiner CA, Jiranek WA, Berry DJ. Prevalence of Total Hip and Knee Replacement in the United States. J Bone Joint Surg Am. 2015 Sep 2;97(17):1386-97. doi: 10.2106/JBJS.N.01141. PMID 26333733
- [Background] Moerman S, Mathijssen NMC, Tuinebreijer WE, Vochteloo AJH, Nelissen RGHH. Hemiarthroplasty and total hip arthroplasty in 30,830 patients with hip fractures: data from the Dutch Arthroplasty Register on revision and risk factors for revision. Acta Orthop. 2018 Oct;89(5):509-514. doi: 10.1080/17453674.2018.1499069. Epub 2018 Aug 6. PMID 30080985
- [Background] Tangsataporn S, Safir OA, Vincent AD, Abdelbary H, Gross AE, Kuzyk PR. Risk Factors for Subsidence of a Modular Tapered Femoral Stem Used for Revision Total Hip Arthroplasty. J Arthroplasty. 2015 Jun;30(6):1030-4. doi: 10.1016/j.arth.2015.01.009. Epub 2015 Jan 21. PMID 25701193

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: 124
Groups:
- SAGITTA EVL R: Patients of this group have received a total hip replacement with a SAGITTA EVL R Stem.
Period: Overall Study
Arm/Group | SAGITTA EVL R
Started | 120; 124 124 (Number of unit is corresponding to : Operated Hips)
Completed | 71; 73 124 (Number of unit is corresponding to : Operated Hips)
Not Completed | 49; 51 124
Not completed — Death | 46
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | SAGITTA EVL R
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex information were not collected for one subject
  Participants
    number analyzed (Participants) | 119
    Female | 64
    Male | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: Kilograms] | 77.5 (20.7)

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate of Stems
Time Frame: at 5 years follow-up
Population: Patient that have reached the last Follow-up.
Measure: Number; unit: Percentage of stem unrevised
Units Other Than Participants: Stems implanted
Arm/Group | SAGITTA EVL R
Number analyzed (Participants) | 71
Number analyzed (Stems implanted) | 73
Percentage of stem unrevised | 94

2. Secondary Outcome: Patient Satisfaction
Description: The information will be collected from the patient by answering a Yes/No question at last follow-up. The following result correspond to the number of patients that have been satisfied
Time Frame: at 5 years follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SAGITTA EVL R
Number analyzed (Participants) | 71
Participants | 53

3. Secondary Outcome: Functional Improvement
Description: The information will be collected from both the patient through questionnaires to compare preoperatively situtation to last follow-up situtation. The patient will estimate the improvement in 3 scales: improved/unchanged/Worsen.
  The result present number of patient answering improved.
Time Frame: at 5 years follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SAGITTA EVL R
Number analyzed (Participants) | 71
Participants | 41

4. Secondary Outcome: Pain Release
Description: The information will be collected from both the patient through questionnaires to compare preoperatively situtation to last follow-up situtation. The patient will estimate the pain diminution with 2 options: Yes or No diminution of pain. Result presents the number of patient having pain diminution
Time Frame: at 5 years follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SAGITTA EVL R
Number analyzed (Participants) | 71
Participants | 53

ADVERSE EVENTS:
Time Frame: At 5 years follow-up
Description: [Not specified]
Arm/Group | SAGITTA EVL R
All-Cause Mortality (participants affected / at risk) | 46/120
Serious Adverse Events (participants affected / at risk) | 0/120
Other Adverse Events (participants affected / at risk) | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT05153473/Prot_000.pdf